CLINICAL TRIAL: NCT01814007
Title: Safety Evaluation of Multiple CoolSculpting Treatments
Brief Title: Multiple CoolSculpting Treatment Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zeltiq Aesthetics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ZA13-001
Record Dates: First submitted 2013-03-04; First posted 2013-03-19 (Estimated); Results first posted 2020-12-02 (Actual); Last update posted 2021-05-17 (Actual); Status verified 2020-11

CONDITIONS: Body Fat Disorder
Keywords: Lipolysis; Cryolipolysis; Fat Reduction
MeSH Terms: interventions — Lipectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- CoolSculpting Treatment Group (Experimental): CoolSculpting treatments will be performed on all subjects with 1 cooling cycle on the lower abdomen, plus simultaneous treatment of both flanks, one cooling cycle each. Two control units will be utilized at protocol-defined temperatures and durations.
  Interventions: Device: The Zeltiq CoolSculpting System

INTERVENTIONS:
Device: The Zeltiq CoolSculpting System — Non-invasive cooling is applied to the treatment area with a defined cooling rate and duration.
  Other Names: Cryolipolysis; Lipolysis

SUMMARY:
To evaluate the safety of same-day CoolSculpting treatments and to assess the impact on serum lipids and liver-related tests.

DETAILED DESCRIPTION:
The study will evaluate the safety of multiple same-day CoolSculpting treatments and will assess any impact on serum lips or liver-related analytes,

ELIGIBILITY:
Inclusion Criteria

* Male or female subjects > 18 years of age.
* Subject who has been assessed to receive multiple CoolSculpting treatments on the abdomen and flanks, defined as follows:

  1. Lower Abdomen - One 60 minute cycle with CoolMax,
  2. Right and Left Flank - One 60 minute cycle per flank, with CoolCurve+ or CoolCore, simultaneously.
* Subject has not had weight change exceeding 10 pounds in the preceding month.
* Subject with body mass index (BMI) up to 30. BMI is defined as weight in pounds multiplied by 703 divided by the square of the height in inches.
* Subject agrees to not making any major changes in their diet or lifestyle during the course of the study.
* Subject has read and signed a written informed consent form.

Exclusion Criteria

* Subject has had an invasive (e.g., liposuction, mesotherapy, abdominoplasty) or non-invasive fat reduction and/or body contouring procedure in the area of intended treatment within the past 6 months.
* Subject needs to administer, or has a known history of subcutaneous injections into the area of intended treatment (e.g., heparin, insulin) within the past month.
* Subject has a known history of cryoglobulinemia, cold urticaria, or paroxysmal cold hemoglobinuria.
* Subject has a history of hernia in the area(s) to be treated.
* Subject is pregnant or intending to become pregnant during the study period (in the next 4 months).
* Subject is lactating or has been lactating during the past 3 months.
* Subject is unable or unwilling to comply with the study requirements, such as blood draw.
* Subject is currently enrolled in a clinical study of any other unapproved investigational drug or device.
* Subject has a history of lipodosis or other confounding metabolic diseases.
* Subject is taking or has taken medication within the past 3 months which may affect the metabolic function.
* Patient has a history of diabetes.
* Any other condition or laboratory value that would, in the professional opinion of the investigator, potentially affect the subject's response or the integrity of the data or would pose an unacceptable risk to the subject.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2013-03; Primary Completion 2013-07-22 (Actual); Study Completion 2013-10-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Bachelor, MD, Principal Investigator — Innovation Research Center
Locations (3):
- United States (3):
  - Innovation Research Center, Pleasanton, California
  - Ed Becker, MD, Walnut Creek, California
  - Bowes Dermatology Group, Miami, Florida

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Multiple same day cryolipolysis treatments for the reduction of subcutaneous fat are safe and do not affect serum lipid levels or liver function tests — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC5573959/

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment Group: All study subjects are treated on the abdomen and flanks with the Zeltiq System: Non-invasive cooling is applied to the treatment area with a defined cooling rate and duration.
Period: Overall Study
Arm/Group | Treatment Group
Started | 35
Completed | 34
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Groups:
- Treatment Group: All study subjects are treated on the abdomen with the Zeltiq System: Non-invasive cooling is applied to the treatment area with a defined cooling rate and duration.
Arm/Group | Treatment Group
Number analyzed (Participants) | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.2 (2.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 8
Region of Enrollment [Number; unit: participants]
  United States | 35

OUTCOME MEASURES:

1. Primary Outcome: Evaluation of Liver- Related Tests Over Time
Description: Blood draws will be collected pre-treatment, 1-week, 4-weeks, 12-weeks post treatment. Changes in each analyte was evaluated for consistency with normal variation and for change relative to the reference range of the component (high/low), pre-treatment versus post-treatment by an independent physician. The independent physician reviewer was provided with laboratory results and other pertinent information for each subject, including demographic, medical history, and concomitant medications. For every change in laboratory value over time, the reviewer was required to make a determination of whether the change in value represented a clinically meaningful change. In addition, for any change in a laboratory value that exceeded 25% change, or any value outside of normal range, the reviewer was required to provide a written rationale for the determination of clinical meaningfulness.
Time Frame: Pre-treatment; 1 week, 4 weeks, and 12 weeks post-treatment
Population: Blood draws completed on 35 subjects at baseline. Two liver-related test results unavailable for 1 subject at baseline. Blood draws at the 1 week, 4 week and 12 week time periods reflect 34 subjects as one of the 35 subjects enrolled withdrew from the study. Liver-related test values were analyzed for each time point.
Measure: Least Squares Mean (Standard Deviation); unit: units per liter (U/L)
Groups:
- CoolSculpting Treatment Group: CoolSculpting of Abdomen and Flanks
  The Zeltiq CoolSculpting System: Non-invasive cooling is applied to the treatment area with a defined cooling rate and duration.
Arm/Group | CoolSculpting Treatment Group
Number analyzed (Participants) | 35
units per liter (U/L)
  Baseline Alk Phosphatase: number analyzed (Participants) | 34
  Baseline Alk Phosphatase | 62.12 (15.72)
  1 week post treatment Alk Phosphatase: number analyzed (Participants) | 34
  1 week post treatment Alk Phosphatase | 63.88 (14.71)
  4 weeks post treatment Alk Phosphatase: number analyzed (Participants) | 34
  4 weeks post treatment Alk Phosphatase | 63.74 (15.61)
  12 week post treatment Alk Phosphatase: number analyzed (Participants) | 34
  12 week post treatment Alk Phosphatase | 62.06 (15.4)
  Baseline AST-SGOT | 19.66 (5.16)
  1 week post treatment AST-SGOT: number analyzed (Participants) | 34
  1 week post treatment AST-SGOT | 19.76 (6.93)
  4 weeks post treatment AST-SGOT: number analyzed (Participants) | 34
  4 weeks post treatment AST-SGOT | 22.15 (8.77)
  12 week post treatment AST-SGOT: number analyzed (Participants) | 34
  12 week post treatment AST-SGOT | 23.03 (16.33)
  ALT-SGPT Baseline: number analyzed (Participants) | 34
  ALT-SGPT Baseline | 17.68 (7.48)
  ALT-SGPT 1 week post treatment: number analyzed (Participants) | 34
  ALT-SGPT 1 week post treatment | 20.44 (12.4)
  ALT-SGPT 4 weeks post treatment: number analyzed (Participants) | 34
  ALT-SGPT 4 weeks post treatment | 20 (10.57)
  ALT-SGPT 12 weeks post treatment: number analyzed (Participants) | 34
  ALT-SGPT 12 weeks post treatment | 19.35 (15.27)

2. Primary Outcome: Evaluation of Liver-Related Tests Over Time
Description: Blood draws will be collected pre-treatment, 1-week, 4-weeks, 12-weeks post treatment. Changes in each analyte was evaluated for consistency with normal variation and for change relative to the reference range of the component (high/low), pre-treatment versus post-treatment by an independent physician. The independent physician reviewer was provided with laboratory results and other pertinent information for each subject, including demographic, medical history, and concomitant medications. For every change in laboratory values over time, the reviewer was required to make a determination of whether the change in value represented a clinically meaningful change. In addition, for any change in a laboratory value that exceeded 25% change, or any value outside of normal range, the reviewer was required to provide a written rationale for the determination of clinical meaningfulness.
Time Frame: Pretreatment, 1 week, 4 weeks 12 weeks post-treatment
Population: Total bilirubin test results were not available for 2 subjects for the baseline visit. Of the 35 subjects enrolled in the study, 1 subject withdrew from the study and had no further blood draws.
Measure: Least Squares Mean (Standard Deviation); unit: mg/dl
Arm/Group | Treatment Group
Number analyzed (Participants) | 35
mg/dl
  Total Bilirubin Baseline: number analyzed (Participants) | 33
  Total Bilirubin Baseline | 0.65 (0.36)
  Total Bilirubin 1 week: number analyzed (Participants) | 34
  Total Bilirubin 1 week | 0.53 (0.24)
  Total Bilirubin 4 weeks: number analyzed (Participants) | 34
  Total Bilirubin 4 weeks | 0.61 (0.27)
  Total Bilirubin 12 weeks: number analyzed (Participants) | 34
  Total Bilirubin 12 weeks | 0.58 (0.28)

3. Primary Outcome: Evaluation of Serum Lipid Values Over Time
Description: as for outcome 2
Time Frame: Pre-treatment, 1 week, 4 weeks, 12 weeks post-treatment
Population: Of the 35 subjects enrolled, 1 subject withdrew and did not have blood draws performed after the baseline visit.
Measure: Least Squares Mean (Standard Deviation); unit: mg/dl
Arm/Group | Treatment Group
Number analyzed (Participants) | 35
mg/dl
  Cholesterol Baseline | 186.54 (39.08)
  Cholesterol 1 week: number analyzed (Participants) | 34
  Cholesterol 1 week | 185.62 (36.9)
  Cholesterol 4 weeks: number analyzed (Participants) | 34
  Cholesterol 4 weeks | 188.38 (37.6)
  Cholesterol 12 weeks: number analyzed (Participants) | 34
  Cholesterol 12 weeks | 189.18 (39.76)
  Triglycerides Baseline | 76.97 (32.49)
  Triglycerides 1 week: number analyzed (Participants) | 34
  Triglycerides 1 week | 80.53 (33.19)
  Triglycerides 4 weeks: number analyzed (Participants) | 34
  Triglycerides 4 weeks | 77.68 (33.22)
  Triglycerides 12 weeks: number analyzed (Participants) | 34
  Triglycerides 12 weeks | 83.35 (38.59)
  HDL Cholesterol Baseline | 71.03 (26.83)
  HDL Cholesterol 1 week: number analyzed (Participants) | 34
  HDL Cholesterol 1 week | 68.56 (26.35)
  HDL Cholesterol 4 weeks: number analyzed (Participants) | 34
  HDL Cholesterol 4 weeks | 70.59 (27.36)
  HDL Cholesterol 12 weeks: number analyzed (Participants) | 34
  HDL Cholesterol 12 weeks | 73.79 (31.69)
  LDL Cholesterol Baseline | 99.97 (23.12)
  LDL Cholesterol 1 week: number analyzed (Participants) | 34
  LDL Cholesterol 1 week | 100.94 (26.78)
  LDL Cholesterol 4 weeks post treatment: number analyzed (Participants) | 34
  LDL Cholesterol 4 weeks post treatment | 102.65 (21.73)
  LDL Cholesterol 12 weeks post treatment: number analyzed (Participants) | 34
  LDL Cholesterol 12 weeks post treatment | 102.5 (28.72)
  VLDL Cholesterol Baseline | 15.67 (6.83)
  VLDL Cholesterol 1 week: number analyzed (Participants) | 34
  VLDL Cholesterol 1 week | 16.12 (6.5)
  VLDL Cholesterol 4 weeks post treatment: number analyzed (Participants) | 34
  VLDL Cholesterol 4 weeks post treatment | 15.45 (6.62)
  VLDL Cholesterol 12 weeks post treatment: number analyzed (Participants) | 34
  VLDL Cholesterol 12 weeks post treatment | 16.8 (7.85)

4. Primary Outcome: Safety of the Device and/or Procedure as Assessed by the Incidence of SAE and UADE
Description: The primary safety end point is the incidence of Serious Adverse Events (SAE) and Unanticipated Adverse Device Effects (UADE).
Time Frame: 12 weeks post treatment
Population: All treated subjects were included in the safety analysis population.
Measure: Number; unit: participants
Arm/Group | CoolSculpting Treatment Group
Number analyzed (Participants) | 35
participants
  Serious AE reported | 1
  UADEs reported | 0

5. Secondary Outcome: Safety as Evaluated by the Number and Severity of All Reported Adverse Events.
Description: All adverse will be assessed for frequency and severity from the time of enrollment though the 12 week follow-up visit.
Time Frame: 12 weeks post-treatment
Population: All subjects treated with the CoolSculpting device were included in the analysis population.
Measure: Count of Participants; unit: Participants
Arm/Group | CoolSculpting Treatment Group
Number analyzed (Participants) | 35
Participants
  Moderate severity AE | 1
  Mild severity AE | 2

6. Secondary Outcome: Pain: Assessment of Pain Scores Reported on the Day of Treatment and at 12 Weeks Post-treatment.
Description: Pain scores are collected using a 0 (no pain) to 10 (worst possible pain) scale. Scores will be collected immediately post-treatment and at the 12 week follow-up visit.
Time Frame: Treatment day and 12 week post-treatment follow-up
Population: All subjects treated with the CoolSculpting System were included in the analysis population. One (1) subject was withdrawn from the study by the investigator after treatment, therefore pain scores reflect 35 subjects analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CoolSculpting Treatment Group
Number analyzed (Participants) | 35
score on a scale
  Post Treatment Pain Score | 4 (3)
  12-week Pain Score: number analyzed (Participants) | 34
  12-week Pain Score | 0 (0)

7. Secondary Outcome: Side Effects in Treatment Area
Description: Clinical assessments of the skin at the treatment sites to be performed immediately post-treatment, and at the 12 week follow-up visit. Subjects will be evaluated for skin changes at the treatment sites. The scale used by clinicians for the assessments is 0 = absent, 1= minor, 2= moderate, 3= severe.
Time Frame: Treatment day and 12 week post-treatment follow-up
Population: The analysis population included all subjects treated with the CoolSculpting System. 1 subject did not complete the final follow-up visit. The abdomen, left and right flanks were clinically assessed immediately post treatment and at 12 weeks. At 12 weeks, 102 treatment sites were assessed.
Measure: Number; unit: Treatment sites
Units Other Than Participants: Treatment sites
Arm/Group | CoolSculpting Treatment Group
Number analyzed (Participants) | 35
Number analyzed (Treatment sites) | 103
Treatment sites
  Bruising absent immed post treatment | 64
  Minor bruising immed post treatment | 31
  Moderate bruising immed post treatment | 7
  Severe bruising immed post treatment | 1
  Erythema absent immed post treatment | 0
  Minor erythema immed post treatment | 54
  Moderate erythema immed post treatment | 46
  Severe erythema immed post treatment | 3
  Edema absent immed post treatment | 31
  Minor edema immed post treatment | 46
  Moderate edema immed post treatment | 25
  Severe edema immed post treatment | 1
  Numbness absent immed post treatment | 14
  Minor numbness immed post treatment | 30
  Moderate numbness immed post treatment | 47
  Severe numbness immed post treatment | 12
  Tingling absent immed post treatment | 56
  Minor tingling immed post treatment | 32
  Moderate tingling immed post treatment | 12
  Severe tingling immed post treatment | 3
  Other skin effect immed post treatment | 1
  Bruising absent at 12 wks: number analyzed (Participants) | 34
  Bruising absent at 12 wks: number analyzed (Treatment sites) | 102
  Bruising absent at 12 wks | 102
  Erythema absent at 12 weeks: number analyzed (Participants) | 34
  Erythema absent at 12 weeks: number analyzed (Treatment sites) | 102
  Erythema absent at 12 weeks | 102
  Edema absent at 12 weeks: number analyzed (Participants) | 34
  Edema absent at 12 weeks: number analyzed (Treatment sites) | 102
  Edema absent at 12 weeks | 102
  Numbness absent at 12 weeks: number analyzed (Participants) | 34
  Numbness absent at 12 weeks: number analyzed (Treatment sites) | 102
  Numbness absent at 12 weeks | 102
  Tingling absent at 12 weeks: number analyzed (Participants) | 34
  Tingling absent at 12 weeks: number analyzed (Treatment sites) | 102
  Tingling absent at 12 weeks | 102
  Other skin effect absent at 12 weeks at 12 weeks: number analyzed (Participants) | 34
  Other skin effect absent at 12 weeks at 12 weeks: number analyzed (Treatment sites) | 102
  Other skin effect absent at 12 weeks at 12 weeks | 102

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from the time of enrollment through the 12-week follow-up visit.
Description: Adverse events (AE) will be assessed continuously throughout the study. An adverse event is defined as any untoward medical occurrence in a subject, regardless of whether the event is related to the device. UADE = Any serious adverse effect on health and safety or any life-threatening problem or death caused by, or associated with a device.
Groups:
- CoolSculpting Treatment Group: All subjects treated with the CoolSculpting System are included in the CoolSculpting Treatment Group.
Arm/Group | CoolSculpting Treatment Group
All-Cause Mortality (participants affected / at risk) | 0/35
Serious Adverse Events (participants affected / at risk) | 1/35
Other Adverse Events (participants affected / at risk) | 2/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CoolSculpting Treatment Group (N=35)
Inguinal hernia repair (Gastrointestinal disorders) | 1 (1) — The subject reported an inguinal hernia to the site. Surgery was performed to repair the injury; the subject was discharged on the surgery day. Investigator determined the hernia was not related to the CoolSculpting device or procedure.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CoolSculpting Treatment Group (N=35)
Liver related test results out of normal range (Hepatobiliary disorders) | 1 (1) — Blood draw performed at12 week time point showed elevation in ALT-SGOT and ALT-SGPT. Moderate ETOH consumption the night prior to the test was reported. The blood draw was repeated 2 months following. ALT-SGOT and ALT-SGPT were within normal limits.
Bronchitis (Infections and infestations) | 1 (1) — Subject reported fever and cough and was diagnosed with bronchitis. Antibiotics and nasal spray were prescribed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No